CLINICAL TRIAL: NCT02361931
Title: Prospective, Multicenter, Single-blind, Randomized, Controlled Clinical Trial on Safety and Efficacy of a Novel Topical Formulation Containing Erythropoietin for the Treatment of Diabetic Foot Ulcers
Brief Title: Topical Erythropoietin Hydrogel Formulation for Diabetic Foot Ulcers
Acronym: Remede d'Or
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Remedor Biomed Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0252-12-RMB
Record Dates: First submitted 2012-08-12; First posted 2015-02-12 (Estimated); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Diabetic Foot Ulcer
Keywords: erythropoietin; diabetic chronic wounds; wound healing; chronic wounds; topical treatment; re-epithelization; inflammation
MeSH Terms: conditions — Diabetic Foot; Inflammation | interventions — Standard of Care; Hydrogels

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment group (erythropoietin) (Experimental): 10 patients receive RMD-G1 (gel with 2000 IU/ml of erythropoietin) as an adjunct therapy to standard of care (SOC). Topical application on wound bed, daily for 12 weeks.
  Interventions: Drug: A hydrogel containing erythropoietin
- Control group (standard of care) (Placebo Comparator): 10 patients receive SOC alone daily for 12 weeks. A moisturizing gel is applied on wound bed as a part of SOC.
  Interventions: Drug: Hydrogel (as a part of SOC)

INTERVENTIONS:
Drug: A hydrogel containing erythropoietin — Standard of wound care, which includes initial debridement, wound cleansing, pressure relief, and infection control. RMD-G1 applied daily onto a clean wound at 0.25g per sq.cm. of wound surface. After its application, the wound is covered with a dressing in order to prevent leakage of the gel and contamination of the wound area.
  Other Names: Standard of care (SOC)
  Arms: Treatment group (erythropoietin)
Drug: Hydrogel (as a part of SOC) — Standard of wound care, which includes initial debridement, wound cleansing, pressure relief, and infection control. Hydrogel applied daily onto a clean wound at 0.25g per sq.cm. of wound surface. After its application, the wound is covered with a dressing in order to prevent leakage of the gel and contamination of the wound area.
  Other Names: Standard of care (SOC)
  Arms: Control group (standard of care)

SUMMARY:
Remedor has developed a patented technology (RMD-G1), which comprises erythropoietin (EPO) as the active pharmaceutical ingredient (API) in a carbopol-based hydrogel with an FN matrix. RMD-G1 was designed to maintain EPO stability and activity over long periods and to optimize the administration of EPO onto the wound bed.

RMD-G1 is indicated for treating DFUs in adult patients with diabetes mellitus and aims to accelerate the healing of diabetic foot ulcers. RMD-G1 is an adjunct treatment, and not a substitute for good diabetic wound care, which includes initial debridement, wound cleansing, pressure relief, and infection control. In this trial, RMD-G1 is applied daily onto a clean wound at 0.25g per sq. cm. wound surface. After its application, the wound will be covered with a dressing in order to prevent leakage of the hydrogel and contamination of the wound area.

DETAILED DESCRIPTION:
Delayed healing of a neuroischaemic diabetic foot ulcer (DFU) has been related to prolonged local inflammatory response, an unstable provisional matrix, increased degradation of the extracellular matrix, lack of growth factors and their receptors that are crucial for healing, fibroblast dysfunction, impaired neovascularization, increased oxidative stress, and cellular apoptosis in the wound bed, all of which collectively hinder re-epithelialisation and wound closure.

Erythropoietin (EPO) is an approved drug which is widely used for treating anaemia. EPO is a well-known glycoprotein hormone, which is primarily produced by the tubular cells of the kidney. EPO is widely known for regulating the red blood cell mass by stimulating differentiation and proliferation of precursor cells and hindering apoptosis of erythroid cells in the bone marrow. Millions of people have received EPO since its market approval by the US Food and Drug Administration in 1989 as a treatment of anaemia in patients with chronic kidney disease and later on as a treatment for chemotherapy-associated anaemia. There is growing evidence that both systemic administration and topical EPO application to skin wounds in animals with experimentally-induced diabetes mellitus (DM) and in patients with DM accelerates the healing of these wounds. This accelerated wound healing is mediated by EPO because it concomitantly suppresses the inflammatory response and apoptosis and stimulates angiogenesis, re-epithelialization, and collagen deposition.

Growing studies in experimental healthy and diabetic animals have demonstrated that systemic or topical treatment with EPO onto acute and chronic wounds and burns is safe and effective. Recently, the molecular mechanisms of EPO action in wound repair have been elucidated. EPO acts on all cutaneous cells that are involved in the wound healing process by promoting cellular differentiation and proliferation, exerting cytoprotective actions, and inhibiting inflammation and apoptosis due to the presence of EPO receptors in these cells [Hamed et al. 2014].

The aim of this multicenter, single-blind, randomized, controlled clinical trial is to evaluate the safety and efficacy of topical RMD-G1 treatment for DFUs. This study is an exploratory proof-of-concept study on RMD-G1 treatment for DFU.

ELIGIBILITY:
Inclusion Criteria:

Patients must satisfy all of the following inclusion criteria to be included in the study:

1. Male or female over the age of 18;
2. Diabetes Mellitus type 2;
3. Have a single non-infected Diabetic Hard-to-Heal wound (ulcers/foot ulcers), Wagner grade I or II documented for at least 4 weeks that has not shown signs of healing despite standard treatment;
4. 2 sq.cm. ≤ Wound area at start of treatment ≤ 10 sq.cm.;
5. At least moderate blood perfusion into the affected limb as defined by Ankle Brachial Index (ABI) of >0.4 or if ABI >1.3 then toe pressure > 50 mmHg;
6. Undergo a current physical examination, which reveals no clinically significant abnormalities, except diabetes or diabetic ulcer/wound related condition;
7. Be available for the entire study period, and be able and willing to adhere to protocol requirements;
8. Provide written informed consent prior to admission into the study;
9. no surgical revascularization of the limb with the DFU was done in the previous two months.

Exclusion Criteria:

Patients will be excluded from the study if they meet any of the following exclusion criteria:

1. Diabetes Mellitus non Type 2;
2. Have a glycosylated haemoglobin (HbA1c) >10.0%;
3. Have a body mass index (BMI) > 40 Kg/m2;
4. Have visible bone exposure at wound site;
5. Subjects whose study ulcer size decreases by more than 30% during this initial standard-of-care phase (pre-treatment phase);
6. Have any signs of infection in the wound (which could be linked to raised body temperature), abscess, cellulitis, necrosis, erythema, mild drainage or known osteomyelitis;
7. Have a history of HIV or a clinically significant cardiac, gastrointestinal, endocrine, neurological, liver, or kidney disease;
8. Anemia (Hemoglobin < 9 g/dL) or White Blood Cells count > 11,000/μL or Platelets count < 100,000/μL or liver function tests > 3 times upper normal lab values or Creatinine > 3 mg/dL; any indication of malnourishment (Albumin < 3 g/dL); INR>2 or any other clinically significant blood and urinalysis tests per the physician's discretion
9. Have any clinically significant chronic or acute illness during the 4 weeks prior to admission into the study, except diabetes type2 or during screening period;
10. Patients on concomitant medications that alter blood glucose levels (e.g. ACE inhibitors, lipid lowering agents, etc.) who have not been on a stable dosage regimen for at least 4 weeks prior to entry into the study and who cannot maintain a stable dosage throughout the study;
11. Malignant disease except Basal Cell Carcinoma or Cervical Carcinoma in situ; Chemotherapy treatment or severely immunosuppressed for any reason that would limit or preclude healing in the opinion of the Investigator;
12. Females who are pregnant, lactating, of child-bearing potential, or post-menopausal for less than 2 years, not using a medically approved method of contraception (i.e., oral, transdermal, or implanted contraceptives, intrauterine device, diaphragm, condom, abstinence, or surgical sterility), or females who test positive on a blood-based pregnancy test;
13. Participation in a clinical study or use of an investigational drug within 30 days prior to admission to this study;
14. Residing in a nursing facility and/or are bed-ridden (unable to come to receive treatment at the clinic).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-03-21 (Actual); Primary Completion 2018-06-11 (Actual); Study Completion 2018-06-12 (Actual)

PRIMARY OUTCOMES:
Number of participants without adverse events following RMD-G1 treatment | 24 weeks
  Absence of serious adverse events associated with the RMD-G1 treatment.
Number of participants with the reduction of wound area by 75%$ or more | 12 weeks
  Wound area will be assessed weekly for 75% closure or more of the wound area, which is defined as 75% epithelialization of the wound with no secretions.

SECONDARY OUTCOMES:
Number of patients with hypersensitivity at the wound site. | 12 weeks
  Weekly assessments of wound site for signs of hypersensitivity to the RMD-G1 treatment.
Speed of healing | 12 weeks
  The time to reach complete wound closure (days).
Reduction of wound area | 12 weeks
  Absolute wound area regression (AWAR) (cm2) will be assessed weekly.
Partial wound closure | 4 weeks
  The number of participants with a wound surface area regression ≥ 50% and ≥ 75% by week 4.
Rate of wound closure | 12 weeks
  Mean rate of wound closure (sq. cm./day) will be assessed weekly.
Recurrence of closed wounds | 24 weeks
  Number of wound recurrence cases

CONTACTS AND LOCATIONS:
Overall Officials: Yehuda Ullman, Professor, Study Chair — Rambam Health Care Campus
Locations (5):
- Israel (5):
  - HaEmek Medical Center, Afula
  - Rambam Health Care Campus, Haifa
  - Edith Wolfson Medical Center, Holon
  - Galilee Medical Center, Nahariya
  - Poriya Medical Center (a.k.a. Baruch Padeh Medical Center), Tiberias

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hamed S, Ullmann Y, Belokopytov M, Shoufani A, Kabha H, Masri S, Feldbrin Z, Kogan L, Kruchevsky D, Najjar R, Liu PY, Kerihuel JC, Akita S, Teot L. Topical Erythropoietin Accelerates Wound Closure in Patients with Diabetic Foot Ulcers: A Prospective, Multicenter, Single-Blind, Randomized, Controlled Trial. Rejuvenation Res. 2021 Aug;24(4):251-261. doi: 10.1089/rej.2020.2397. Epub 2021 Apr 1. PMID 33504262